CLINICAL TRIAL: NCT04315740
Title: THE ULTRAFINE PROJECT - A Study of Acute Health Effects of Exposure to Particles Generated by Candles and Cooking
Brief Title: Acute Health Effects Due to Ultrafine Particles From Candles and Cooking
Acronym: Ultrafine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Torben Sigsgaard, Professor, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 191100
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-03

CONDITIONS: Candle Burning; Cooking; Lung Function Decreased; DNA Damage; Subjective Health; Asthma
Keywords: Particle contamination; Indoor air; Acute health effects; RCT; Asthma
MeSH Terms: conditions — Respiratory Insufficiency; Asthma | interventions — Environment, Controlled

STUDY DESIGN:
Intervention Model Description: A randomised double-blinded crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The exposure was generated in small adjacent chamber and thereby led into the exposure chamber using a pipe connection and a small negative pressure. Thus, the exposure could not be observed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clean Air (Sham Comparator): Just clean air - no exposure
  Interventions: Other: Clean Air
- Cooking (Experimental): Four ovens were frying pork - one at a time. When the first oven finished, the next oven started and so forth for approx. 7 hours.
  Interventions: Other: Particles from cooking
- Candles (Experimental): 10 lit candles were placed at a table. Burning for approx. 7 hours with light ventilation.
  Interventions: Other: Particles from candles

INTERVENTIONS:
Other: Particles from candles — Generating fine and ultrafine particles from lit candles
  Arms: Candles
Other: Particles from cooking — Generating fine and ultrafine particles from frying pork in an oven
  Arms: Cooking
Other: Clean Air — Nothing but clean air
  Arms: Clean Air

SUMMARY:
People spend up to 90% of their life indoor, and the way we live and behave in our homes has substantial effects on our health and well-being. Particle contamination is suggested to have substantial negative effects on health, with candles and cooking emitting the largest amount of particles, thus being the largest contributors to indoor air pollution.

The overall aim of the present project is to contribute to increased understanding of the association between indoor particulate air pollution and health and well-being.

DETAILED DESCRIPTION:
Introduction: People spend up to 90% of their life indoor, and the way we live and behave in our homes has substantial effects on our health and well-being. Particle contamination is suggested to have substantial negative effects on health, with candles and cooking emitting the largest amount of particles, thus being the largest contributors to indoor air pollution. Little is known about the potential adverse health effects of candles and cooking, and people with asthma may be more susceptible.

Aim: To investigate local and systemic effects of short-term exposure to lit candles and cooking among young asthmatics.

Design: In a randomised double-blinded cross-over study non-smoking asthmatics (18-25 years) were exposed for five hours at three different exposure conditions separated by 14 days; A) clean filtered air, B) lit candles and C) cooking emissions under controlled environmental conditions.

Measurements: TSI P-TRAK Ultrafine Particle Counter was used for particle counts. Health effects, including lung function (FEV1/FVC) and fraction of exhaled nitric oxide (FeNO) were evaluated in relation to local and systemic effects prior to, right after and 24 h. after exposure.

Analysis: Mixed methods approach taking both time and exposure into account.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-25
* Medically treated / physician diagnosed mild seasonal asthma
* Never smoker or ex-smoker ≥ 6 months
* Allergy > 1 common allergy

Exclusion Criteria:

* Any other disease that could influence the study parameters
* Conditions that prevent safe access to the climate chambers (such as claustrophobia)
* Perennial asthma
* Need for continuous medical treatment for asthma
* Pregnancy

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Particles in Exhaled Air (Surfactant Protein A & Albumin) | Time Frame: At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  PExA: Subjects performed repeated breath maneuvers allowing for airway closure and re-opening, and exhaled particles were optically counted and collected on a membrane using the (novel) PExA® instrument set-up.

SECONDARY OUTCOMES:
Change in Lung Function (FEV1 & FVC) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Spirometry
Change in Fractional exhaled nitric oxide (FENO) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  NIOX VERO system; Aerocrine AB, Sweden
Change in Blood samples | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Cytokines (IL-8), DNA-damages
Change in nasal volume (using Acoustic rhinometry) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Is used to assess the nasal cross sectional area and volume. The left and right nasal cavity were studied alternatively until three reproducible measurements were obtained. The minimum cross sectional cavity area was calculated from the means of the measurements. By integration of the area-distance curve, the sum of the volume 2 to 4 (vol2-4) from the nostril was determined on both sides.
Change in biomarkers in Saliva Sample | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  An oral svap from Salivette was placed in the mouth of the participant to collect saliva by gently chewing the swab for one minute. Afterwards the saturated swab was removed to the suspended insert and closed firmly with a lid. Then the sample was transferred to a freezer and stored for -80 C until further analysis. The sample will be analyzed for biomarkers (amylase, cortisol, substance P, lysozyme and secretory IgA.)
Change in Subjective Symptoms | Every 30 minute during 5 hours of exposure
  In the exposure chamber participants were asked to fill out a symptom questionnaire every 30 minute regarding their well-being and experienced symptoms in eyes, nose and throat. The participants were asked to score their evaluation (rate the strength) of symptoms by placing a cross on a 130 mm open Visual Analogue Scale (VAS). The intensity of any discomfort was registered as the length in mm from the left of the scale to the marker. The scores were rated from 0 to 100% with highest number corresponding to highest discomfort. Health effects were evaluated in relation to rated changes in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Laursen, MSc, Principal Investigator — Department of Public Health, Aarhus Universitet
Locations (1):
- Climate Chambers, Dept. Public Health, Aarhus University, Aarhus, Central Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No